CLINICAL TRIAL: NCT05777993
Title: A Rollover Study to Provide Continued Access to Mitapivat for Participants Who Previously Completed an Agios-Sponsored Mitapivat Study
Brief Title: A Study to Provide Continued Access to Mitapivat for Participants Who Previously Completed an Agios-Sponsored Mitapivat Study
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-025
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pyruvate Kinase Deficiency; Anemia, Hemolytic
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia, Hemolytic | interventions — mitapivat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mitapivat (Experimental): Participants will receive mitapivat of 5, 20 or 50 milligrams (mg), orally, twice daily (BID), based on the last dose received by the participants in the antecedent study. Mitapivat will be administered from Day 1 up to end of treatment period of this study.
  Interventions: Drug: Mitapivat

INTERVENTIONS:
Drug: Mitapivat — Tablets
  Other Names: AG-348; Mitapivat sulfate; PYRUKYND®

SUMMARY:
The purpose of this study is to provide continued access to mitapivat for participants who completed an Agios-sponsored mitapivat study (antecedent) and do not have commercial access to mitapivat.

DETAILED DESCRIPTION:
Participants will continue the mitapivat dose regimen that they were receiving at the final visit of their antecedent study.

ELIGIBILITY:
Inclusion Criteria:

* Has completed an Agios-sponsored adult pyruvate kinase (PK) deficiency study of mitapivat within 1 day of enrollment in this rollover study;
* Is unable to obtain mitapivat treatment due to country regulations or lack of commercial access;
* Was deriving clinical benefit from mitapivat treatment at the completion of the antecedent study, in the opinion of the Investigator;
* For women of childbearing potential, must be abstinent of sexual activities that may result in pregnancy as part of their usual lifestyle or agree to use 2 forms of contraception, 1 of which must be considered highly effective, from the time of providing informed consent, throughout the study, and for 28 days after the last dose of study drug. The second form of contraception can be an acceptable barrier method;
* Written informed consent from the participant before any study-related procedures are conducted and willing to comply with all study procedures for the duration of the study;
* Agrees not to participate in other interventional clinical studies, including other studies of mitapivat, during participation in this study.

Exclusion Criteria:

* Has discontinued treatment with mitapivat before completing the antecedent study;
* Known allergy or other contraindication to mitapivat or its inactive ingredients (microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, mannitol, Opadry II Blue [hypromellose, titanium dioxide, lactose monohydrate, triacetin, and FD&C Blue #2]);
* Any medical, hematologic, psychological, or behavioral condition(s) or prior or current therapy that, in the opinion of the Investigator, may confer an unacceptable risk to participating in the study also excluded are:

  * Participants who are institutionalized by regulatory or court order
  * Participants with any condition(s) that could create undue influence (including but not limited to incarceration, involuntary psychiatric confinement, and financial or familial affiliation with the Investigator or Sponsor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 6.2 years
Percentage of Participants With AEs and SAEs, Graded by Severity | Up to approximately 6.2 years
  The severity of all AEs will be graded by the Investigator according to Version 4.03 of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) on a 5-point severity scale (Grade 1 through Grade 5) where Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening and Grade 5 is fatal.
Percentage of Participants With AEs Considered by the Investigator to be Related to Study Drug | Up to approximately 6.2 years
Percentage of Participants With SAEs Considered by the Investigator to be Related to Study Drug | Up to approximately 6.2 years

CONTACTS AND LOCATIONS:
Locations (4):
- McMaster Centre for Transfusion Medicine McMaster University, Hamilton, Ontario, Canada
- Japan (3):
  - Tohoku University Hospital, Sendai, Miyagi
  - Kyoto Katsura Hospital, Kyoto
  - Toho University - Omori Medical Center, Ōta-ku

IPD SHARING:
Plan to Share IPD: No